CLINICAL TRIAL: NCT02206438
Title: The Clinical Efficacy of Supraglottic Airway Device, Self-pressurized Air-Q Intubating Laryngeal Airway (ILA -SP) in Adult Patients: Comparison With Classic-laryngeal Airway (c-LMA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 3-2014-0081
Record Dates: First submitted 2014-07-28; First posted 2014-08-01 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2016-10

CONDITIONS: Surgery
Keywords: supraglottic airway devices; the classic laryngeal mask airway; the self-pressurised air-Q intubating laryngeal airway in adult patients; elective surgery of short duration (less than 2 hr) undergoing general anesthesia using supraglottic airway in adult patients

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1)C-LMA group (Experimental)
  Interventions: Device: Insertion of C-LMA
- 2)Air-Q group (Active Comparator)
  Interventions: Device: Insertion of air-Q according

INTERVENTIONS:
Device: Insertion of C-LMA — After induction of general anesthesia, C-LMA or Air-Q was inserted according to randomly allocated group.
  Arms: 1)C-LMA group
Device: Insertion of air-Q according — After induction of general anesthesia, C-LMA or Air-Q was inserted according to randomly allocated group.
  Arms: 2)Air-Q group

SUMMARY:
Supraglottic airway devices (SADs) are well established in anesthetic practice. Among these devices ,classic laryngeal airway has been typically widely used. The self-pressurised air-Q (air-Q) is newly developed supraglottic airway devices. It is a new single-use device that may optimise the airway sealing while reducing the potential for postoperative complications such as sore throat. The overall structure of the air-Q SP is identical to the original air-Q, except with regard to the inflatable cuff. The aim of this randomized trial was to compare the clinical performance of the classic LMA and the air-Q SP.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (20-75 of age) scheduled for elective surgery of short duration (less than 2 hr) undergoing general anesthesia using supraglottic airway

Exclusion Criteria:

* Patients with a potentially difficult airway, risk of aspiration such as gastroesophageal reflux disease, or active upper respiratory tract infection

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
airway leak pressure measured after device insertion | within 5min to 10 min insertion of each device
  Airway leak pressure was determined by adjusting the expiratory valve of the breathing circle to 40 cmH2O (fixed fresh gas flow 3 L/min) and recording the pressure when equilibrium was reached.

SECONDARY OUTCOMES:
Insertion time | During and 1 min after insertion of each device
  Insertion time was defined as the time from the attending anesthesiologist picking up the LMA until the confirmation on capnography.

OTHER OUTCOMES:
Ease of insertion | During and 1 min after insertion of each device
  Ease of insertion was graded from 1 to 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Human research Protection Center, Gangnam Severance Hospital,, Seoul, South Korea

REFERENCES:
- [Derived] Ha SH, Kim MS, Suh J, Lee JS. Self-pressurized air-Q(R) intubating laryngeal airway versus the LMA(R) Classic: a randomized clinical trial. Can J Anaesth. 2018 May;65(5):543-550. doi: 10.1007/s12630-018-1082-6. Epub 2018 Feb 6. PMID 29524199